CLINICAL TRIAL: NCT05502133
Title: Identification of Acute Intermittent Porphyria Modifying Genes
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Robert Desnick, Dean for Genetics and Genomic Medicine Emeritus, Professor and Chair Emeritus, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 18-1800
Record Dates: First submitted 2022-08-04; First posted 2022-08-16 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Acute Intermittent Porphyria (AIP)
MeSH Terms: conditions — Porphyria, Acute Intermittent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Acute Intermittent Porphyria (AIP): Symptomatic patients with Acute Intermittent Porphyria (AIP)
  A member of an AIP family who possesses an AIP pathogenic mutation and is/has been symptomatic (experienced acute attacks). Parents with no known HMBS mutations or heterozygote with familial mutation or a first, second or third degree relative of the above.

SUMMARY:
This study proposes to identify the predisposing/protective modifying genes that underlie the acute attacks in symptomatic patients with Acute Intermittent Porphyria (AIP), an autosomal dominant inborn error of heme biosynthesis.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent
* 12 years of age or older
* Willingness to provide blood/saliva and urine samples, and clinical information
* A member of an AIP family, defined as (must meet one of the following):

  1. proband: possesses an AIP pathogenic mutation and is/has been symptomatic (experienced acute attacks in the opinion of the investigator)
  2. Parents (no known HMBS mutations or heterozygote with familial mutation)
  3. First, second, or third degree relative of (a) or (b)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A member of an AIP family who possesses an AIP pathogenic mutation and is/has been symptomatic (experienced acute attacks). Parents with no known HMBS mutations or heterozygote with familial mutation or a first, second or third degree relative of the above.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Odds ratios (OR) of the effects of identified modifier genes/variants | Day 1
  There are no primary and secondary endpoints. This is an exploratory genetic study.
  Exploratory Endpoints: Odds ratios (OR) of the effects of identified modifier genes/variants.
  (If putative predisposing or protective gene variants are identified)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Desnick, Ph.D, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Not feasible.